CLINICAL TRIAL: NCT04274231
Title: Integrative Genomic Analysis Reveals Cancer-associated Gene Mutations in Chronic Myeloid Leukemia Patients With Tyrosine Kinase Inhibitor Resistance or Intolerance
Brief Title: Cancer-associated Gene Mutations in CML Treatment With TKIs by NGS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, xuna, doctor, Nanfang Hospital, Southern Medical University
Other Study IDs: CML-NGS
Record Dates: First submitted 2020-02-16; First posted 2020-02-18 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Different Gene Between Different TKIs Effection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TKI best effect group: TKI best effect was defined achieve complete cytogenetic response (CCyR)after 3 months of treatment and the level of BCR/ABL<10% after 3 months of treatment,the level of BCR/ABL<1% .
  Interventions: Genetic: different effection
- TKI resistance group: TKI resistance was defined as the lack of a complete hematologic response (CHR) after 3 months of TKI treatment, the lack of any cytogenetic response after 6 months of treatment, the lack of major cytogenetic response (MCyR) (Ph-positive cells > 35%) after 12 months of treatment, an increase of white blood cell (WBC) count in at least two consecutive samplings (with a doubling of the count from the nadir to ≥ 20×109/L or an absolute increase of ≥ 50×109/L), or a relapse after a CHR or MCyR.
  Interventions: Genetic: different effection
- TKI intolerance group: TKI intolerance was defined as at least grade 3 nonhematologic toxicity or grade 4 hematologic toxicity persisting for more than 7 days, related to TKIs at any dose.
  Interventions: Genetic: different effection

INTERVENTIONS:
Genetic: different effection — Analysis of the reasons for treatment

SUMMARY:
We performed targeted-capture sequencing of 127 known and putative cancer-related genes of patients who best effect to TKIs ,or intolerance to TKIs,or resistance to TKIs by next-generation sequencing (NGS) .

ELIGIBILITY:
Inclusion Criteria:

1. Chronic myeloid leukemia-Chronic phase(CML-CP) patients treated with receiveTyrosine kinase inhibitor -TKI(including imatinib, dasatinib and nilotinib) for more than 1 years
2. best effect to TKIs ,or intolerance to TKIs,or resistance to TKIs according to Q-pcr detected BCR/ABL(IS) in peripheral blood and hematologic response and cytogenetic response
3. Informed consent of the patient or his legal representative

Exclusion Criteria:

1. Patients had history of CML-AP or CML-BC
2. CML Patients who have received allogeneic hematopoietic stem cell transplantation
3. CML Patients who have received immunotherapy (except interferon, including car-t and other cellular immunotherapy)
4. Woman who is pregnant or nursing

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Best effect to TKI group Intolerance to TKI group Resistance to TKI group
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-16 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
cancer-associated gene mutations in CML treatment with TKIs by NGS | 1 year after TKI treatment
  We performed targeted-capture sequencing of 127 known and putative cancer-related genes of patients who best effect to TKIs ,or intolerance to TKIs,or resistance to TKIs by next-generation sequencing (NGS)

CONTACTS AND LOCATIONS:
Overall Officials: H Nanfang, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- NanfangH, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes